CLINICAL TRIAL: NCT03948269
Title: Internet- and Mobile-based Group Treatment of Menopausal and Psychological Health of Chinese Women: a Study Protocol for a Randomized Non-inferiority Trial
Brief Title: The Effect of Internet- and Mobile-based Group Treatment in Menopausal Women
Acronym: IMGTMP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Southeast University, China (Other)
Collaborators: The Affiliated Obstetrics and Gynecology Hospital of Nanjing Medical University (Unknown)
Responsible Party: Principal Investigator, Dan Li, Principal investigator, Southeast University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Southeast Menopausal Protocol
Record Dates: First submitted 2019-05-09; First posted 2019-05-13 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Menopausal Syndrome
Keywords: menopause; group treatment; mood swing; quality of life

STUDY DESIGN:
Intervention Model Description: Mixed-effects models (random intercept) with interaction effects of group and time will be conducted on primary and secondary repeating outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet- and mobile-based group treatment (Experimental): the therapy consists of 10 modules (15 hours in total) in groups of 8 participants each over a period of 10 weeks and one follow-up meeting (2 hours) 12 weeks after the 10th module (week 22). Each module is adapted from the previous literature on CBT rationale and will be conducted online on WeChat, a mobile social networking software with 1 billion users in 2018. First, we will establish a WeChat group containing the imGT group members and psychiatrists, in which everyone can talk instantly. The interactive treatments will be conducted every Friday evening for a duration of 1.5 hours via text, audio or video messaging.
  Interventions: Behavioral: group behavioral cognitive therapy
- Face-to-face group treatment (Active Comparator): 10 modules will be conducted every weekend in the psychological counseling room of The Affiliated Obstetrics and Gynaecology Hospital of Nanjing Medical University.
  Interventions: Behavioral: group behavioral cognitive therapy

INTERVENTIONS:
Behavioral: group behavioral cognitive therapy — First, we will establish a WeChat group containing the imGT group members and psychiatrists, in which everyone can talk instantly. The interactive treatments will be conducted every Friday evening for a duration of 1.5 hours via text, audio or video messaging. Table 1 summarizes the module topics and provides detailed information on the treatment program. All modules will be saved for repeated viewing after completion. Second, we will establish another WeChat program named Punched-in which participants report on aspects of their everyday life such as diet, sports, readings or mood, according to the plan made by psychiatrists, via text, audio, photo or video message. This program will only be visible to and able to be commented on by participants and psychiatrists.

SUMMARY:
Background: Menopause syndrome generally occurs with and is related to psychological problems. However, Internet- and mobile-based group treatment (imGT) may improve women's physiological and psychological conditions.

Objective: To investigate the efficacy of group treatment with or without Internet- and mobile-based treatment of menopause, mood swings and quality of life status.

Methods: This protocol is for a randomized controlled clinical trial with a sample of 144 menopausal women divided into 2 groups: imGT and face-to-face group treatment (ffGT). The primary outcome will be the menopausal symptom improvement of the two groups, as assessed by Greene Climacteric Scale. The secondary outcomes will be quality of life, assessed by the Short Form 36 Health Survey Questionnaire; insomnia, assessed by the Pittsburgh Sleep Quality Inventory; anxiety, assessed by the Hamilton Anxiety Rating Scale; and therapeutic alliance, assessed by the Working Alliance Inventory-Short Revised. imGT will be performed once a week for 1.5 hours for 10 weeks with a daily Punched-in on the WeChat App; ffGT will be performed once a week for 1.5 hours for 10 weeks. All outcomes will be assessed at baseline, at a post-intervention evaluation (week 10), and at a follow-up evaluation (week 22).

Discussion: This study will be the first clinical trial to examine the effects of imGT on menopausal women in China. If imGT is found to be equivalent to or superior to ffGT, it will facilitate easier access to menopausal health services, which may be feasible to offer to other medical institution.

ELIGIBILITY:
Inclusion Criteria:

* aged 40~60, in menopausal transition or post-menopause, according to the STRAW +10 definition
* have Internet access
* have mobile phone access
* have sufficient knowledge of the Chinese language
* have scored in the clinical range for menopause syndrome from the psychiatric interview
* have signed a consent form that will be provided to eligible participants.

Exclusion Criteria:

* not completing informed consent
* presence of any of the following diseases: hyperthyroidism, coronary atherosclerotic heart disease, hypertension (BP≥140/90 mmHg), pheochromocytoma, neurasthenia, psychosis, or other diseases closely related to the main disease
* troublesome drinking
* drug use (hypnotics or hormone therapy) in the past 14 days, which might affect mood.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
Greene Climacteric Scale | week 0
  Greene Climacteric Scale is used for evaluating menopausal symptoms. It contains 21 questions covering 5 domains: anxiety, depression, somatic symptoms, vasomotor symptoms, and sexual function. Each question is answered on a 4-point Likert scale. The answers to all 21 questions are summed to give a total quality-of-life measure; a higher score indicates a worse quality of life. According to the hypothesis and PRO-specific domains of this trial, vasomotor symptoms, anxiety and depression will be analysed specifically. The Chinese version of this questionnaire has a high validation (0.90), and the Cronbach's alpha coefficient is 0.95, while its test-retest reliability is 0.94 (P <0.01).
Greene Climacteric Scale | week 10
  Menopause symptoms after 10 sessions of group cognitive behavioral therapy
Greene Climacteric Scale | week 22
  Menopause symptoms of one follow-up meeting

SECONDARY OUTCOMES:
The Short Form 36 Health Survey Questionnaire | week 0
  The Short Form 36 Health Survey Questionnaire (SF36) is widely used for evaluating the potential benefits of healthcare interventions. It is comprised of eight dimensions (including physical functioning, social functioning, role limitations, mental health, energy/vitality, pain, general health perceptions), and the score ranges from 0 to 100, where better health achieves higher scores. This questionnaire was chosen because of the validation of the Chinese version with a sensitivity of 0.72~0.88 and specificity of 87.5%~100%.
The Short Form 36 Health Survey Questionnaire | week 10
  Quality of life
The Short Form 36 Health Survey Questionnaire | week 22
  Quality of life
Pittsburgh Sleep Quality Index | week 0
  The Pittsburgh Sleep Quality Index (PSQI) is a self-rating inventory that evaluates sleep quality and disturbances within a 4-week time interval. It comprises 19 individual items with a global score ranging from 0 to 21. The correlation coefficient of PSQI for t-test reliability was 0.87. A Chinese PSQI score >7 yielded a sensitivity of 98.3% and specificity of 90.2% in distinguishing between good and poor sleepers (kappa= 0.89, p<0.01)
Pittsburgh Sleep Quality Index | week 10
  Insomnia
Pittsburgh Sleep Quality Index | week 22
  Insomnia
The Hamilton Anxiety Rating Scale | week 0, 10, 22
  The Hamilton Anxiety Rating Scale (HAM-A) is a rating scale developed to measure the symptoms of anxiety neurosis. It is a semi-structured clinician-rated interview consisting of 14 items that measure both psychological anxiety and somatic anxiety. A 5-point scale ranging from 0 (not present) to 4 (severe) is used, where the total severity score is 0-56; <17 indicates mild anxiety and 25-30 is considered moderate-severe. The Chinese version of HAM-A will be used in this study.
The Hamilton Anxiety Rating Scale | week 10
  Anxiety
The Hamilton Anxiety Rating Scale | week 22
  Anxiety
The Working Alliance Inventory-Short Revised | week 0, 10
  The Working Alliance Inventory-Short Revised (WAI-SR) provides an assessment of the therapeutic alliance and contains 12 items with three dimensions of working alliance: agreement on the tasks of therapy, agreement on the goals of therapy and development of an affective bond between client and therapist. Items are rated on a 5-point scale (range from 1= "never" to 5= "always").
The Working Alliance Inventory-Short Revised | week 10
  Therapeutic alliance
Client Satisfaction Qestionnaire-8 (CSQ-8) | week 10
  Treatment satisfaction will be measured by the Client Satisfaction Qestionnaire-8 (CSQ-8), which evaluates the service utilization and psychotherapy outcome measures with high internal consistency (coefficient α = .91).

CONTACTS AND LOCATIONS:
Overall Officials: Jing Ms Kong, Master, Principal Investigator — the Affiliated Obstetrics and Gynaecology Hospital of Nanjing Medical University
Locations (1):
- the Affiliated Obstetrics and Gynaecology Hospital of Nanjing Medical University, Nanjing, Jiangsu, China